CLINICAL TRIAL: NCT00305734
Title: Phase II Trial of PS-341 (Bortezomib, NSC-681239) Followed by the Addition of Gemcitabine at Progression in Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: Bortezomib and Gemcitabine in Treating Patients With Recurrent or Metastatic Nasopharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02690; SWOG-S0506; U10CA032102 (NIH); CDR0000462635 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Nasopharyngeal Cancer; Stage IV Nasopharyngeal Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Bortezomib; Gemcitabine

ARMS (1):
- Treatment (bortezomib, gemcitabine hydrochloride) (Experimental): Patients receive bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a CR receive 2 additional courses of treatment with bortezomib.
  Patients who experience disease progression on single-agent bortezomib and did not receive prior gemcitabine hydrochloride may begin combination therapy within 10-28 days of the last dose of bortezomib. Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and bortezomib IV on days 1, 4, 8, 11. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a CR receive 2 additional courses beyond the confirmed CR.
  Interventions: Drug: bortezomib; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving bortezomib together with gemcitabine works in treating patients with recurrent or metastatic nasopharyngeal cancer. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with gemcitabine may kill more tumor cells

DETAILED DESCRIPTION:
OBJECTIVES: Primary I. Assess the response probability (confirmed and unconfirmed, complete and partial responses) and 3-month progression-free survival rate in patients with metastatic or recurrent nasopharyngeal carcinoma (NPC) who are treated with bortezomib.

Secondary I. Estimate 1-year progression-free survival and assess quantitative toxicities in this group of patients treated with bortezomib.

II. Evaluate the response probability (confirmed and unconfirmed, complete and partial) in the subset of patients who progress on bortezomib, with measurable disease at the time of progression, and go on to receive bortezomib and gemcitabine hydrochloride combination therapy.

III. Estimate 1-year overall survival of all patients treated with this regimen.

IV. Estimate 6-month progression-free survival from the start of combination therapy and assess quantitative toxicities in the subset of patients who progress on bortezomib and receive combination therapy.

V. Explore, in a preliminary manner, the relationship between changes in Epstein-Barr virus DNA level, NF-kB DNA-binding activity, and methylation status of E-cadherin promoter with clinical outcomes.

OUTLINE: This is a multicenter study of bortezomib.

Patients receive bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 additional courses of treatment with bortezomib.

Patients who experience disease progression on single-agent bortezomib and did not receive prior gemcitabine hydrochloride may begin combination therapy within 10-28 days of the last dose of bortezomib. Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and bortezomib IV on days 1, 4, 8, 11. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a CR receive 2 additional courses beyond the confirmed CR.

After the completion of study treatment, patients are followed periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed nasopharyngeal carcinoma (NPC) of one of the following subtypes:

  * Non-keratinizing (WHO type II)
  * Undifferentiated (WHO type III)
* Disease meets one of the following stage criteria:

  * Stage IVC at diagnosis
  * Persisted, metastasized, or recurred after definitive surgery, radiotherapy, and/or chemotherapy
* Measurable disease

  * If only measurable disease is within a prior radiation therapy port, disease progression must be clearly demonstrated
* No known CNS metastases
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN) OR creatinine clearance ≥ 60 mL/min
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin normal
* SGOT or SGPT ≤ 2.5 times ULN
* Zubrod performance status 0-2
* No peripheral neuropathy > grade 1
* No prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the patient has been disease-free for 5 years
* Not pregnant or nursing
* Fertile patients must use effective contraception
* More than 6 months since prior myocardial infarction
* No New York Heart Association class III or IV cardiac problems
* No uncontrolled angina
* No severe uncontrolled ventricular arrhythmias
* No acute ischemia by ECG
* No active conduction system abnormalities
* No known hypersensitivity to bortezomib, boron, or mannitol
* See Disease Characteristics
* No prior therapy with gemcitabine hydrochloride, bortezomib, or other proteasome inhibitors

  * No more than 28 days since discontinuation of single-agent bortezomib
  * Patients with prior gemcitabine hydrochloride treatment are eligible for single-agent bortezomib treatment but NOT for combination treatment
* No more than one prior chemotherapy regimen for the treatment of metastatic or recurrent NPC

  * At least 28 days since prior treatment and recovered
* At least 24 weeks since prior adjuvant chemotherapy
* At least 24 weeks since prior chemotherapy as a radiosensitizer for initial locally advanced disease
* At least 28 days since prior radiotherapy and recovered
* At least 28 days since prior surgery and recovered
* No other concurrent therapy for NPC, including any of the following:

  * Radiotherapy
  * Chemotherapy
  * Immunotherapy
  * Biologic therapy
  * Other investigational drugs
  * Gene therapy
* No colony-stimulating factor therapy during the first course of study therapy
* No concurrent highly active antiretroviral therapy (HAART) in HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-08; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Objective response rate (confirmed and unconfirmed, complete and partial response) based on the Response Evaluation Criteria in Solid Tumors (RECIST) in patients treated with bortezomib | Up to 3 years
Progression-free survival rate | 3 months

SECONDARY OUTCOMES:
Response probability (confirmed and unconfirmed, complete and partial response) based on the RECIST in patients treated with bortezomib and gemcitabine hydrochloride | Up to 3 years
Progression-free survival rate | 6 months
Progression-free survival rate | 1 year
Adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 | Up to 3 years
  95% confidence intervals will be estimated.
Overall survival | 1 year
Relationship between Epstein-Barr virus (EBV) deoxyribonucleic acid (DNA) level, NF-kB DNA- binding activity, and methylation status of E-cadherin promoter with clinical outcome | Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Shibata, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States